CLINICAL TRIAL: NCT03622879
Title: Effect of Mirror Therapy with Cutaneous Electrical Sensory Stimulation on Lower Limb Motor Functions in People with Stroke: a Single-blinded Randomized Controlled Trial
Brief Title: Mirror Therapy with Cutaneous Electrical Sensory Stimulation on Lower Limb Motor Functions in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018_GRF_NG
Record Dates: First submitted 2018-07-10; First posted 2018-08-09 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Mirror therapy; Transcutaneous Electric Nerve Stimulation; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- MT + TENS (Experimental): The subject will adopt a semi-seated position on a bed while the mirror board is positioned between the legs perpendicular to the subject's midline. The paretic leg will be positioned behind the mirror, with the intact leg facing the reflective surface. All subjects will be reminded to focus on the image in the mirror during MT training. All subjects will receive concurrent TENS stimulation over the common peroneal nerve while practising bilateral lower limb exercises. After 15 minutes of priming with TENS + MT, all subjects will perform 60 minutes of lower limb task-oriented training.
  Interventions: Behavioral: MT; Device: TENS; Behavioral: Lower-limb task-oriented training
- Placebo-MT+TENS (Placebo Comparator): In the Placebo-MT+TENS group, the experimental set-up and protocol will be the same as in the MT+TENS group, except that the reflecting surface of the angle-adjustable mirror was covered with paper. After 15 minutes of priming, all subjects will perform 60 minutes of lower limb task-oriented training.
  Interventions: Device: TENS; Behavioral: Lower-limb task-oriented training
- MT+placebo-TENS (Placebo Comparator): In the MT+placebo-TENS group, the experimental set-up and protocol will be the same as in the MT+TENS group. The only difference is that placebo stimulation will be applied to the paretic limb from identical-looking TENS devices with the electrical circuit disconnected inside. After 15 minutes of priming, all subjects will perform 60 minutes of lower limb task-oriented training.
  Interventions: Behavioral: MT; Behavioral: Lower-limb task-oriented training
- control training (Sham Comparator): All subjects will perform 60 minutes of lower limb task-oriented training only.
  Interventions: Behavioral: Lower-limb task-oriented training

INTERVENTIONS:
Behavioral: MT — A customised angle-adjustable frame with a mirror board (60 × 90 cm) will be used. All subjects are instructed to perform hip flexion/abduction, knee flexion/extension and ankle dorsiflexion/plantarflexion on the intact-limb during a 15 minutes period.
  Arms: MT + TENS; MT+placebo-TENS
Device: TENS — TENS will be delivered to the common peroneal nerve of the paretic leg. The stimulation frequency will be 100Hz and with an intensity just below the motor threshold.
  Arms: MT + TENS; Placebo-MT+TENS
Behavioral: Lower-limb task-oriented training — The lower-limb task-oriented training comprises 6 exercises, namely stepping up and down, heel lift a dorsiflexed position, partial squatting, kicking a ball with alternate legs, gait re-education and transition training. Each exercise last for 10 minutes

SUMMARY:
This study aims to evaluate the effectiveness of concurrent mirror therapy (MT) and transcutaneous electrical nerve stimulation (TENS) in augmenting the efficacy of the lower limb task-oriented training in people with stroke. It is hypothesize that MT combined with TENS would be superior to sham-mirror therapy with TENS, or MT with placebo-TENS, or control training only in improving lower limb motor functions and walking ability in people with stroke when combined with the lower limb task-oriented training.

DETAILED DESCRIPTION:
The application of transcutaneous electrical nerve stimulation (TENS) over a paretic lower limb could augment the effects of task-oriented exercise therapy on lower limb motor function in people with stroke, possibly through increased excitability of sensorimotor cortex.

In mirror therapy (MT), the intact limb performs motor tasks while its mirror reflection is superimposed over the covered paretic limb, creating a visual illusion of enhanced function over the paretic limb. The visual input during MT could substitute for reduced proprioceptive inputs and increase spatial attention of the paretic limb, which could improve motor function of the paretic limb, possibly through increased cortical activity in the lesioned hemisphere and mirror neurone system.

The next question concerns whether MT could be combined with TENS and whether their synergetic effects could maximise the motor output of paretic limbs in people with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. have had a single stroke with ischemic brain injury or intracerebral haemorrhage diagnosed by magnetic resonance imaging or computed tomography within the previous 6 to 36 months;
2. have at least 5 degrees of active ankle dorsiflexion in the antigravity position;
3. are able to walk 10 m independently with or without a walking aid;
4. are able to score 6 or higher out of 10 on the abbreviated mental test;
5. have no unilateral neglect, hemianopia or apraxia;
6. have no skin allergy (e.g. redness or itchiness to the electrical stimulation pads) to electrical stimulation or electrodes; and
7. are able to follow instructions and give informed consent.

Exclusion Criteria:

1. have any additional medical, cardiovascular or orthopaedic condition that would hinder proper treatment or assessment;
2. have visual deficits that may hinder them from benefiting from the mirror visual feedback;
3. have receptive dysphasia; or
4. are involved in drug studies or other clinical trials.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The Change of Fugl-Meyer Assessment of Lower Extremity (FMA-LE) | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  FMA-LE is used to evaluate the lower extremity motor control, including reflexes, voluntary control of isolated movement and coordination. The scale score ranging from 0 to 34, with 17 items and ordinal scoring from 0 to 2. A higher score indicates a better lower extremity motor control. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).

SECONDARY OUTCOMES:
The Change of Paretic ankle dorsiflexor strength | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  The subject's paretic ankle dorsiflexor strength (in kilograms) is measured with a Nicholas hand-held dynamometer (model 01,160, Lafayette Instrument Company, Lafayette, IN) in supine lying position. The muscle strength will be measured twice. The average strength of the 2 trials will be recorded. A higher value indicated a better paretic ankle dorsiflexor strength. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).
The Change of Paretic ankle plantarflexor strength | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  The subject's paretic ankle plantarflexor strength (in kilograms) is measured with a Nicholas hand-held dynamometer (model 01,160, Lafayette Instrument Company, Lafayette, IN) in supine lying position. The average strength of the 2 trials will be recorded. A higher value indicated a better paretic ankle plantarflexor strength. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).
The Change of 10-m walk test | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  10-m walk test is used to measure the walking speed in a short distance. The subject will be asked to walk 10 meter in a normal comfortable speed and maximum speed condition, respectively. The completion time will be records by stopwatch. Each condition will be repeated for 2 times. The completion time will be averaged. The shorter the completion time indicated the better performance in 10-m walk test. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).
The Change of Timed 'Up and Go' test | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  The Time 'Up and Go' test is used to measure the Functional mobility. Each subject will be required to rise from a chair with armrests, walk 3 m forward, turn around, return to the chair and sit down. The time taken to complete this task will be measured in seconds with a stopwatch. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).
The Change of Lower-extremity motor co-ordination test | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  The lower-extremity motor coordination test is used to measure the coordination of both the paretic and intact legs. Two red flat targets will be secured on the floor 30 cm apart. In sitting position with the feet resting flat on the floor and the heels on one of the targets, the participant will be instructed to touch 2 targets alternately with the big toe, as quickly and as accurately as possible, for 20 seconds. The number of times each target is touched will be counted. The more touch times indicated a better performance. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).
The Change of Cantonese version of Community Integration Measures (CIM-C) | Baseline (0 week), Mid-intervention (4 weeks), Post-intervention (8 weeks), 3-month follow-up (20 weeks)
  The level of community integration will be assessed by the Cantonese version of Community Integration Measures (CIM-C). The CIM is a client-centred questionnaire with 10 items; each item rating from 1 to 5 with a total score from 10 to 50. A higher CIM-C score indicates a higher level of community integration. The assessment will be conducted at baseline, mid-intervention (4 weeks), post-intervention (8 weeks) and 3-month follow-up (20 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: SSM Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong